CLINICAL TRIAL: NCT02167399
Title: Evaluation of the Use of the Smart Phone as a Screening and Evaluation Tool to Identify Knee Valgus During Dynamic Activities.
Brief Title: Smart Phone as a Screening and Evaluation Tool to Identify Knee Valgus During Dynamic Activities
Status: Completed | Type: Observational
Sponsor: Mitchell Selhorst (Other)
Responsible Party: Sponsor-Investigator, Mitchell Selhorst, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00222
Record Dates: First submitted 2014-06-10; First posted 2014-06-19 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Leg Injuries
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- smart phone inclinometer: For the smart phone analysis we will be using the tilt meter application which is a digital inclinometer application available on the I phone. The phone will be placed in the vertical position utilizing the bubble level feature of the application. The application will be set to display measurements to the closest tenth of the degree, set to log measurements every 0.2 seconds. The subject will stand with knee extended to 0 degrees and quadriceps muscle activated and upper extremity support on opposite side of stance limb. The phone will be placed in the vertical position on the anterior portion of the middle third of the subject's thigh attached using double sided adhesive tape. Being placed as close as possible to level when attached to the anterior thigh with subject in single limb stance with a reading of less than 1 deg as minimum for correct set-up prior to testing. Immediately prior to testing recording will be initiated logging measurements for later assessment.
- 2-D video analysis: two dimensional video analysis by first placing markers on the subject at the midpoint of the femoral condyles, midpoint of the ankle malleoli, and the proximal thigh along a line from the anterior superior iliac spine (ASIS) to the knee marker. Testing will take place in front of a digital video camera with tape on the floor to give a reference point for the subject being tested. Participants will be tested twice on day 1 and then again 5-9 days later. Subjects will be allowed 2-3 practice trials prior to each test in order to allow the subject to feel comfortable with each test. Following the practice trials the subject will perform 3 trials of each test on bilateral lower extremities. This set up was consistent with the set up by Munro et al.

SUMMARY:
Evidence supports the use of two dimensional video analysis to assess the presence of dynamic knee valgus during generally used screening tasks, however there is limited evidence to support the use of the various smart phone applications as a time and money saving option for clinic use . Subjects that present to the clinic and display dynamic valgus at the knee during the lateral step down test will be given the option to participate in the study. If they consent to the study they will be evaluated with 2-Dimensional video analysis to determine the amount of valgus present at the knee during the lateral step down test. The subject will also have the smart phone attached to their lower leg and the amount of valgus will be concurrently measured by the selected application. The primary objective of this study is to determine the validity of an application on the smart phone to provide an objective measure of dynamic knee valgus. The secondary objective of this study is to determine the possibility of the use of the application as a source of feedback during neuromuscular re-education training in order to decrease or eliminate a subject's dynamic valgus collapse and subsequently decreased their risk for future injury.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* ability to perform a single leg squat, drop jump, and single leg drop without pain

Exclusion Criteria:

* lower extremity injury within 6 months prior to testing
* history of lower extremity surgery
* lower extremity weight bearing restrictions
* inability to follow directions
* neoprene/latex allergy
* Adhesive allergy
* Current neurological or developmental condition
* inability to attend follow-up session
* actively receiving Physical Therapy intervention for varus/valgus impairment
* Current pregnancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: physical therapy clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Agreement in Dynamic lower extremity valgus angles during single leg squat | Baseline
  Patient's dynamic lower extremity valgus during single leg squat will be measured using both 2-D video analysis and smart phone inclinometer analysis. Measurements of 2-D and smart phone will be taken at the same time. Analysis will be repeated at 2nd visit to assess the reliability of the measurements

SECONDARY OUTCOMES:
Agreement in Dynamic lower extremity valgus angles during drop jump | Baseline
  Patient's dynamic lower extremity valgus during a drop jump from a 12 inch step will be measured using both 2-D video analysis and smart phone inclinometer analysis. Measurements of 2-D and smart phone will be taken at the same time. Analysis will be repeated at 2nd visit to assess the reliability of the measurements

OTHER OUTCOMES:
Agreement in Dynamic lower extremity valgus angles during single leg landing drop jump | Baseline
  Patient's dynamic lower extremity valgus during a single leg drop jump from a 12 inch step will be measured using both 2-D video analysis and smart phone inclinometer analysis. Measurements of 2-D and smart phone will be taken at the same time. Analysis will be repeated at 2nd visit to assess the reliability of the measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C Selhorst, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio, United States

REFERENCES:
- [Background] Swenson DM, Collins CL, Fields SK, Comstock RD. Epidemiology of U.S. high school sports-related ligamentous ankle injuries, 2005/06-2010/11. Clin J Sport Med. 2013 May;23(3):190-6. doi: 10.1097/JSM.0b013e31827d21fe. PMID 23328403
- [Background] Munro A, Herrington L, Carolan M. Reliability of 2-dimensional video assessment of frontal-plane dynamic knee valgus during common athletic screening tasks. J Sport Rehabil. 2012 Feb;21(1):7-11. doi: 10.1123/jsr.21.1.7. Epub 2011 Nov 15. PMID 22104115